CLINICAL TRIAL: NCT06951425
Title: A Phase l, Open-Label, Dose-escalation Study to Evaluate the Safety, Tolerability and Antitumor Activity of TH027 CAR-T Cells (TH-CART-027) in Subjects With Relapsed or Refractory Solid Tumors
Brief Title: An Exploratory Clinical Study of the Efficiency and Safety of TH027 in the Treatment of Relapsed/Refractory Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: ThinkingBiomed (Unknown)
Responsible Party: Principal Investigator, Aibin Liang, Professor, Chief Physician, Vice President of Tongji Hospital, Tongji University School of Medicine etc., Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH027-ST001
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of B7H3+ solid tumors (Experimental): Intraperitoneal Infusion for Ovarian Cancer and Peritoneal Metastatic Tumors; Intravenous Infusion for Other Types of Solid Tumors
  Interventions: Drug: TH-CART-027

INTERVENTIONS:
Drug: TH-CART-027 — 3+3 dose escalation design: Dose Level 1: 0.3×10^6 CAR+ T cells /kg; Dose Level 2: 1.0×10^6 CAR+ T cells /kg; Dose Level 3: 3.0×10^6 CAR+ T cells /kg

SUMMARY:
This is a Phase l, Open-Label, Dose-escalation Study to Evaluate the Safety, Tolerabilityand Antitumor Activity of TH027 CAR-T Cell lnjection (TH-CART-027) in Subjects With Relapsed or Refractory Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.The patients were aged from 18 to 75 years old (including the cut-off value), and the gender was not limited;
* 2.The expected survival time was more than 12 weeks;
* 3.ECOG score was 0-2;
* 4.One of the following tumor types was confirmed by pathology: osteosarcoma, neuroblastoma, gastric cancer or lung cancer, and the positive rate of CD276 expression in tumor tissue was more than 30% by immunohistochemistry;
* 5.Patients with ineffective standard treatment methods (such as postoperative recurrence, chemotherapy, radiotherapy, and progression after targeted drugs);
* 6.According to RECIST 1.1, there was at least one measurable lesion (the longest diameter of solid lesion >=10 mm, or the short diameter of lymph node lesion >=15 mm);
* 7.The function of main organs was normal (white blood cell count >= 3 × 10^9 / L, neutrophil count >= 1.5 × 10^9 / L, hemoglobin >= 8.5g/dl, platelet count >= 80 × 10^9 / L and lymphocyte count at 1 × 10^9 / L (including) ~ 4 × 10^9 / L (inclusive);
* 8.The liver and kidney function and cardiopulmonary function meet the following requirements:
* Urea and serum creatinine <= 1.5 × ULN；
* Left ventricular ejection fraction >= 50%;
* Baseline oxygen saturation >= 94%;
* Total bilirubin <= 1.5 × ULN； ALT and AST <= 2.5 × ULN；
* 9.The patient or legal representative can fully understand the significance and risk of this trial and has signed the informed consent.

Exclusion Criteria:

* 1.Patients with history of immune deficiency or autoimmune diseases (including but not limited to rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, insulin-dependent diabetes, etc.); Patients with graft-versus-host disease (GVHD) or need immunosuppressive agents;
* 2.There was a history of other second malignancies in 5 years before screening;
* 3.Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) were positive, and the peripheral blood HBV DNA titer was not within the normal reference value; HCV antibody and HCV RNA in peripheral blood were positive; HIV antibody positive patients; Syphilis was positive;
* 4.Severe heart disease: including but not limited to unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification >= III), severe arrhythmia;
* 5.Unstable systemic diseases judged by researchers: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
* 6.Within 7 days before screening, there were active or uncontrollable infections requiring systemic treatment (except mild urogenital infection and upper respiratory tract infection);
* 7.Pregnant or lactating women, female subjects who plan to conceive within one year after cell transfusion, or male subjects whose partners plan to conceive within one year after cell transfusion;
* 8.Patients who had received CAR-T therapy or other gene modified cell therapy before screening;
* 9.The subjects who were receiving systemic steroid treatment within 7 days before the screening or who needed long-term systemic steroid treatment (except inhalation or local use) were determined by the researchers;
* 10.The ascites increased gradually after 2 weeks of conservative treatment (such as diuresis, sodium restriction, excluding ascites drainage);
* 11.According to the judgment of the researcher, it does not conform to the situation of cell preparation;
* 12.Other researchers think that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety：Incidence of Dose Limiting Toxicity (DLT) | 28 days after the first TH-CART-027 infusion.
  Limiting toxicity type, incidence, and severity of dose limiting toxicities (DLTs) within 28 days after the first TH-CART-027 infusion
Safety：Incidence and severity of adverse events (AEs) | Six months post CAR-T cells infusion.
  To evaluate possible adverse events after TH-CAPT-027 infusion, including the incidence and severity of AEs.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 and 24 months post CAR-T cells infusion.
  Time from treatment initiation to death from any cause.
Objective response rate (ORR) | 3 months post CAR-T cells infusion.
  The assessment will be based on the investigator's evaluation of imaging evaluations, with efficacy evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). ORR refers to the proportion of patients with objective evidence of achieving a Complete Response (CR) or Partial Response (PR). Where applicable, responses recorded after disease progression or initiation of non-investigational anticancer therapy will be excluded.
Progression Free Survival (PFS) | 1 year post CAR-T cells infusion.
  Defined as the time from initiation of the investigational drug to the first occurrence of progressive disease (PD) or death from any cause in the absence of documented PD. If no tumor progression is observed and the subject does not die during the study period, the analysis cutoff date will be determined as the date of the last tumor assessment.
Disease Control Rate (DCR) | 1 year post CAR-T cells infusion
  Defined as the proportion of patients achieving Partial Response (PR), Complete Response (CR), or Stable Disease (SD) according to RECIST 1.1 criteria, relative to the total number of cases in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No